CLINICAL TRIAL: NCT04746235
Title: A Phase 2 Study of Venetoclax in Combination With ASTX727 in Patients With Relapsed/Refractory Acute Myeloid Leukemia, and Newly Diagnosed Elderly Patients With AML Who Are Not Candidates for Intensive Chemotherapy
Brief Title: Venetoclax and ASTX727 for the Treatment of Relapsed, Refractory, or Newly Diagnosed Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1007; NCI-2021-00112 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1007 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-01; First posted 2021-02-09 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — decitabine and cedazuridine drug combination; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine and cedazuridine, venetoclax) (Experimental): Patients receive decitabine and cedazuridine PO daily on days 1-5 and venetoclax PO daily on days 1-28 of the first cycle and on days 1-21 of subsequent cycles. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine and Cedazuridine; Drug: Venetoclax

INTERVENTIONS:
Drug: Decitabine and Cedazuridine — Given PO
  Other Names: ASTX727; CDA Inhibitor E7727/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Combination Agent ASTX727; Cedazuridine/Decitabine Tablet; Inqovi
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies the possible benefits of venetoclax and ASTX727 in treating patients with acute myeloid leukemia that has come back (relapsed) or does not respond to treatment (refractory), or elderly patients with newly diagnosed acute myeloid leukemia who are not candidates for intensive chemotherapy. Venetoclax may help block the formation of growths that may become cancer. ASTX727 is the combination of a fixed dose of 2 drugs, cedazuridine and decitabine. Cedazuridine may slow down how fast decitabine is broken down by the body, and decitabine may block abnormal cells or cancer cells from growing. Giving venetoclax and ASTX727 may help to control the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR) of decitabine and cedazuridine (ASTX727) in combination with venetoclax in patients with refractory/relapsed acute myeloid leukemia (AML).

II. To determine the overall response rate (ORR) of ASTX727 in combination with venetoclax in elderly ((≥ 75 years or ≥ 18 years with comorbidities) patients with newly diagnosed acute myeloid leukemia (AML) not eligible for intensive chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the duration of response, disease-free survival (DFS), and overall survival (OS) of patients with refractory/relapsed AML treated with this combination.

II. To determine similar outcomes for newly diagnosed patients with AML who are not candidates for intensive chemotherapy.

III. To determine the safety of venetoclax in combination with ASTX727 in patients with refractory/ relapsed AML, and newly diagnosed patients with AML not candidates for intensive chemotherapy.

IV. To determine the number of relapsed patients able to proceed to stem cell transplantation upon achieving response with the combination venetoclax/ASTX727 regimen.

EXPLORATORY OBJECTIVE:

I. To characterize the pharmacokinetic (PK) profiles of ASTX727 when combined with venetoclax.

OUTLINE:

Patients receive decitabine and cedazuridine orally (PO) daily on days 1-5 and venetoclax PO daily on days 1-28 of the first cycle and on days 1-21 of subsequent cycles. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients with an objective response are followed every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML by the World Health Organization (WHO) classification who have failed prior therapy, refractory to it or relapsed after prior response. Patients with isolated extramedullary AML are eligible (cohort 1)
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* For cohort 2 (frontline elderly or unfit AML AML), the following inclusion criteria:

  * Confirmed newly diagnosed AML
  * Ineligible for induction therapy defined as

    * Either age >= 75 years
    * Or 18-74 years of age with at least one comorbidity (chronic heart failure [CHF] requiring therapy or eject fraction [EF] =< 50%, carbon monoxide diffusing capability [DLCO] =< 65% or forced expiratory volume in 1 second [FEV1] =< 65%, or ECOG 2 or 3)
    * Creatinine clearance ≥30 mL/min to <45 mL/min
    * Moderate hepatic impairment with total bilirubin >1.5 to ≤3.0 × upper limit of normal (ULN)
* Creatinine clearance ≥ 45 ml/min unless related to the disease (e.g. infiltration)
* Total bilirubin < 2 x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement
* Alanine aminotransferase (ALT) < 3 x ULN unless considered due to leukemic involvement (by biopsy or imaging)
* Able to give written informed consent
* Oral hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and hydroxyurea while the patient is on active study treatment through cycle 1, as needed, for clinical benefit and after discussion with the principal investigator (PI). Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment

Exclusion Criteria:

* Acute promyelocytic leukemia
* Prior therapy with a BCL2 inhibitor
* Symptomatic or uncontrolled CNS leukemia
* Active and uncontrolled comorbidities including active uncontrolled infection, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure New York Heart Association (NYHA) class III/IV, clinically significant and uncontrolled arrhythmia as judged by the treating physician
* Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Within 3 months of treatment initiation
  Will be defined as the proportion of patients who had CR (complete remission), CRp (complete remission with incomplete platelet recovery), CRi (complete remission with incomplete count recovery), PR (partial response) or marrow clearance of blasts within 3 months of treatment initiation among adult patients with acute myeloid leukemia (AML). Response criteria will be modified from the International Working Group for AML. Will estimate the ORR for the combination treatments for each cohort, along with the 90% credible intervals. The association between ORR and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Overall incidence and severity of all adverse events | Up to 5 years post treatment
  Will be assessed by Common Toxicity Criteria version 5.0.

SECONDARY OUTCOMES:
Disease free survival | Up to 5 years post treatment
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Overall survival | Up to 5 years post treatment
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Bazinet A, Garcia-Manero G, Short N, Alvarado Y, Bataller A, Abuasab T, Islam R, Montalbano K, Issa G, Maiti A, Yilmaz M, Jain N, Masarova L, Kornblau S, Jabbour E, Montalban-Bravo G, Rausch CR, Pierce S, DiNardo CD, Kadia T, Daver N, Konopleva M, Huang X, Kantarjian H, Ravandi F. Oral decitabine and cedazuridine plus venetoclax for older or unfit patients with acute myeloid leukaemia: a phase 2 study. Lancet Haematol. 2024 Apr;11(4):e276-e286. doi: 10.1016/S2352-3026(24)00033-4. Epub 2024 Mar 4. PMID 38452788
- See also: M D Anderson Cancer Center — http://www.mdanderson.org